CLINICAL TRIAL: NCT00384332
Title: Orally-Disintegrating vs. Regular Olanzapine Tablets: Effects on Weight and GI Hormones
Brief Title: Medication, Weight Gain and GI Hormones
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Richard C. Shelton, Professor, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 051235
Record Dates: First submitted 2006-10-04; First posted 2006-10-06 (Estimated); Results first posted 2017-07-31 (Actual); Last update posted 2017-07-31 (Actual); Status verified 2017-06

CONDITIONS: Bipolar Depression
Keywords: Bipolar Depression; Weight gain bipolar medicine; side effects olanzapine; gastrointestinal hormones bipolar medicine
MeSH Terms: conditions — Bipolar Disorder | interventions — Olanzapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental): Orally disintegrating olanzapine
  Interventions: Drug: orally-disintegrating olanzapine
- Arm 2 (Experimental): regular olanzapine
  Interventions: Drug: regular olanzapine

INTERVENTIONS:
Drug: orally-disintegrating olanzapine — 5 to 20 mg (daily) orally disintegrating olanzapine for approx.8 weeks.
  Other Names: Zydis
  Arms: Arm 1
Drug: regular olanzapine — 5-20 mg. olanzapine daily for approximately 8 weeks.
  Other Names: Zyprexa
  Arms: Arm 2

SUMMARY:
This is an 8 week study that compares two medications. One medication is olanzapine (5-20 mg daily) whereas the other medication is an orally disintegrating medication. Both medications are used to treat depressed bipolar patients. The main focus of this study is the comparison of these two medications on gastro-intestinal hormones and weight gain.

DETAILED DESCRIPTION:
Olanzapine is undeniably one of the most effective treatments available for all phases of bipolar disorder. After FDA approval for bipolar mania, the drug became one of the most widely prescribed of treatments for this difficult-to-treat disorder. However, concerns about weight gain and the associated metabolic syndrome/type II diabetes have impacted the use of olanzapine.

In fact, weight gain is quite common with olanzapine. For example, in one large scale 8-week placebo-controlled trial of olanzapine in bipolar depression, the olanzapine-treated patients gained an average of 2.59 kg., while placebo patients lost an average of 0.47 kg. Further, weight gain can continue over an extended period of time, mounting to an average of about 6 kg. over one year. It should be noted, however, that in prior studies, no efforts have been made to limit weight gain. More recent data suggest that interventions such as dietary counseling are effective in either preventing or reversing weight gain.

Olanzapine is a potent antagonist of serotonin and histamine 1 receptors. Significant and potentially additive weight gain is associated with blockade of serotonin 2C and Histamine 1 receptors. In addition, serotonin and its receptors are significantly involved in the regulation of gastrointestinal (GI) - related hormone secretion. Animal studies suggest significant involvement of other serotonin receptors in the regulation of appetite, satiety, and GI-related hormones. However, the interplay of selective activation or inhibition of these receptor subtypes is complex, and difficult to distinguish from effects on activity and anxiety. Suffice it to say that activation or blockade of these receptors have differential effects on appetite, satiety, metabolic activity, as well as leptin, secretin, insulin, glucagon, ghrelin, neuropeptide Y, and cholecystokinin.

Weight gain and the corresponding metabolic syndrome represent a "deal killer" with regard to the treatment of most patients. However, one recent small study may be highly relevant to this discussion. De Haan et al. investigated the relative effects of standard olanzapine tablets to the orally-disintegrating form (Zydis) in adolescents and young adults who had gained weight with olanzapine. The group randomly assigned 18 patients to continuation olanzapine tablets or Zydis for a 16-week period. The Zydis-treated patients lost an average of 6.6 kg. while the continuation regular olanzapine group gained 3.7 kg. Although small, this study suggests a potential solution to the weight-gain problem associated with olanzapine.

Most of the pharmacological effects on weight and hormones are thought to be mediated centrally. However, De Haan et al. (de Haan L, et al. Psychopharmacology (Berl). 2004;175:389-390) proposed that at least some of the difference could be attributable to local effects in the GI tract. In particular, the site of absorption was suggested as a possible explanation, with the orally disintegrating form (Zydis) yielding less exposure of the pylorus to olanzapine than the standard Zyprexa tablets.

In this project we will treat 20 patients with bipolar disorder with olanzapine (a widely-used and FDA approved treatment for this condition); patients will be randomly assigned (1:1) to either standard Zyprexa tablets or orally disintegrating Zydis. We will measure symptom improvement and weight gain over the course of the study. Patients will be given dietary counseling prior to initiating either medication. In addition, we will contrast the effects of the treatments on GI-related hormones.

ELIGIBILITY:
Inclusion Criteria:

* A principal diagnosis of bipolar 1 or II disorder
* Ages 18-60
* Physically healthy
* Outpatient status
* Montgomery-Asberg Rating Scale (MADRS) Score greater than or equal to 15
* BMI 23-30
* Able and willing to give written informed consent

Exclusion Criteria:

* Prior history of diabetes (types I or II)
* BMI>30
* Non-fasting blood glucose >124
* Fasting blood glucose >125 or random blood glucose >200
* Presence of dyslipidemia (baseline total cholesterol >240, HDL<50, LDL>160, triglycerides >199)
* Current or past history of a non-affective psychotic disorder
* Alcohol or other substance abuse or dependence in the 6 months prior to the evaluation (except for caffeine)
* Current use of any nicotine products
* Schizoid, schizotypal, or borderline personality disorder
* Treatment with olanzapine in the prior 3 months or any history of non- response to or intolerance of olanzapine or the olanzapine-fluoxetine combination (SymbiaxTM)
* Suicide potential that, in the opinion of the investigator, precludes outpatient treatment or participation in a trial
* Participation of subjects in another drug trial within 30 days of evaluation
* The presence of any current medical condition judged by the investigator to potentially interfere with the study procedures or measures
* The likelihood of requiring hospitalization over the period of the study
* The presence of any clinically-significant laboratory abnormality as judged by the investigator
* Pregnancy or lactation
* History of seizure disorder, excluding febrile seizures of childhood
* Any disorder of taste or smell, including severe nasal allergies
* Any other condition which, in the investigator's judgment might increase the risk to the subject or decrease the chance of obtaining satisfactory data to achieve the objectives of the study
* Being unable to comprehend or follow the study procedures.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2007-01; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard C. Shelton, M.D., Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Background] Tohen M, Vieta E, Calabrese J, Ketter TA, Sachs G, Bowden C, Mitchell PB, Centorrino F, Risser R, Baker RW, Evans AR, Beymer K, Dube S, Tollefson GD, Breier A. Efficacy of olanzapine and olanzapine-fluoxetine combination in the treatment of bipolar I depression. Arch Gen Psychiatry. 2003 Nov;60(11):1079-88. doi: 10.1001/archpsyc.60.11.1079. PMID 14609883
- [Background] Shelton RC. Treating bipolar depression. J Fam Pract. 2003 Mar;Suppl:S14-7. No abstract available. PMID 12676079
- [Background] Farwell WR, Stump TE, Wang J, Tafesse E, L'Italien G, Tierney WM. Weight gain and new onset diabetes associated with olanzapine and risperidone. J Gen Intern Med. 2004 Dec;19(12):1200-5. doi: 10.1111/j.1525-1497.2004.40126.x. PMID 15610330
- [Background] eder-Ischia U, Ebenbichler C, Fleischhacker WW. Olanzapine-induced weight gain and disturbances of lipid and glucose metabolism. Essent Psychopharmacol. 2005;6(2):112-7. PMID 15765795
- [Background] Smith RC, Lindenmayer JP, Bark N, Warner-Cohen J, Vaidhyanathaswamy S, Khandat A. Clozapine, risperidone, olanzapine, and conventional antipsychotic drug effects on glucose, lipids, and leptin in schizophrenic patients. Int J Neuropsychopharmacol. 2005 Jun;8(2):183-94. doi: 10.1017/S1461145705005110. PMID 15737248
- [Background] Cohen D. Diabetes mellitus during olanzapine and quetiapine treatment in Japan. J Clin Psychiatry. 2005 Feb;66(2):265-6; author reply 266-7. doi: 10.4088/jcp.v66n0217b. No abstract available. PMID 15705015
- [Background] Gill SS. Stable monotherapy with clozapine or olanzapine increases the incidence of diabetes mellitus in people with schizophrenia. Evid Based Ment Health. 2005 Feb;8(1):24. doi: 10.1136/ebmh.8.1.24. No abstract available. PMID 15671515
- [Background] Zimmermann U, Kraus T, Himmerich H, Schuld A, Pollmacher T. Epidemiology, implications and mechanisms underlying drug-induced weight gain in psychiatric patients. J Psychiatr Res. 2003 May-Jun;37(3):193-220. doi: 10.1016/s0022-3956(03)00018-9. PMID 12650740
- [Background] Tecott LH, Sun LM, Akana SF, Strack AM, Lowenstein DH, Dallman MF, Julius D. Eating disorder and epilepsy in mice lacking 5-HT2c serotonin receptors. Nature. 1995 Apr 6;374(6522):542-6. doi: 10.1038/374542a0. PMID 7700379
- [Background] Kroeze WK, Hufeisen SJ, Popadak BA, Renock SM, Steinberg S, Ernsberger P, Jayathilake K, Meltzer HY, Roth BL. H1-histamine receptor affinity predicts short-term weight gain for typical and atypical antipsychotic drugs. Neuropsychopharmacology. 2003 Mar;28(3):519-26. doi: 10.1038/sj.npp.1300027. PMID 12629531
- [Derived] Bobo WV, Epstein RA Jr, Shelton RC. Effects of orally disintegrating vs regular olanzapine tablets on body weight, eating behavior, glycemic and lipid indices, and gastrointestinal hormones: a randomized, open comparison in outpatients with bipolar depression. Ann Clin Psychiatry. 2011 Aug;23(3):193-201. PMID 21808751

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants referred by treatment providers.
Groups:
- Arm 1- ODT: Orally disintegrating olanzapine
  orally-disintegrating olanzapine: 5 to 20 mg (daily) orally disintegrating olanzapine for approx.8 weeks.
- Arm 2- SOT: regular olanzapine
  regular olanzapine: 5-20 mg. olanzapine daily for approximately 8 weeks.
Period: Overall Study
Arm/Group | Arm 1- ODT | Arm 2- SOT
Started | 13 | 10
Completed | 9 | 10
Not Completed | 4 | 0
Not completed — Lost to Follow-up | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Total
Number analyzed (Participants) | 13 | 10 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 10 | 23
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Self-reported age.
  years | 36.4 (8.5) | 39.7 (9.9) | 38.05 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 6 | 4 | 10
Region of Enrollment [Number; unit: participants]
  United States | 13 | 10 | 23

OUTCOME MEASURES:

1. Primary Outcome: Weight in Kilograms at Baseline, Weeks 1, 4, 6, and 8
Description: Change in weight from baseline to endpoint in kilograms. Reported as weight in Kilograms at Baseline, Weeks 1, 4, 6, and 8
Time Frame: 10 weeks
Measure: Mean (Standard Error); unit: kilograms
Arm/Group | Arm 1- ODT | Arm 2- SOT
Number analyzed (Participants) | 13 | 10
kilograms
  Baseline | 76.0 (0.6) | 76.1 (0.7)
  Week 1 | 77.4 (0.6) | 77.6 (0.7)
  Week 4 | 77.8 (0.6) | 78.3 (0.7)
  Week 6 | 78.9 (0.7) | 79.4 (0.7)
  Week 8 | 79.1 (0.7) | 80.1 (0.7)

2. Secondary Outcome: Change From Baseline Montgomery Asberg Depression Rating Scale
Description: Montgomery Asberg Depression Rating Scale (MADRS) total score. Construct: Depression severity. Scores below represent mean change scores, endpoint minus baseline. Minimum total score: 0 (no depression). Maximum total score: 60 (severe depression). Lower (more negative) scores indicate a better outcome. There are no subscales.
Time Frame: 10 weeks
Population: Patients with bipolar disorder randomized to orally disintegrating versus regular olanzapine.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 13 | 10
units on a scale | -15.5 (13.1) | -15.5 (13.1)

ADVERSE EVENTS:
Arm/Group | Arm 1- ODT | Arm 2- SOT
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/10
Other Adverse Events (participants affected / at risk) | 5/13 | 6/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1- ODT (N=13) | Arm 2- SOT (N=10)
Increased appetite (Gastrointestinal disorders) | 5 (5) | 6 (6) — Increased appetite

LIMITATIONS AND CAVEATS:
Treatment was not blinded to participants or treating physicians.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No